CLINICAL TRIAL: NCT01974882
Title: Minimizing Post-surgical Pain and Narcotic Administration Through Cryotherapy
Acronym: Ice
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Viraj Master (Other)
Responsible Party: Sponsor-Investigator, Viraj Master, Director of Clinical Research Unit, Emory University
Organization: Emory University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: IRB00004593
Record Dates: First submitted 2013-10-18; First posted 2013-11-04 (Estimated); Last update posted 2013-11-04 (Estimated); Status verified 2013-10

CONDITIONS: Urologic Surgical Procedure
Keywords: abdominal surgery; cryotherapy; pain score; narcotic utilization

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cryotherapy (Experimental): Patients in the cryotherapy study group will have ice packs placed on their abdominal wound for the first hour following surgery.
  Interventions: Other: Ice pack
- Control (No Intervention): No adjunctive therapy following abdominal surgery.

INTERVENTIONS:
Other: Ice pack — Cryotherapy was applied via reusable ice bags filled with ice. Ice packs were immediately applied after the dressing was placed on the wound. The ice pack maintained in place for a continuous 24 hours adn was refilled as needed. After twenty-four hours, patients had the option of using ice packs for as long as they wished. The duration of ice pack usage was noted.
  Arms: Cryotherapy

SUMMARY:
Postoperative pain is an unavoidable consequence of open abdominal surgery. Although cryotherapy, the application of ice to a surgical wound site, has been shown to be effective in reducing postoperative pain in orthopedic, gynecologic, and hernia operations, it has not been assessed in patients who undergo major open abdominal operations. We hypothesized that patients who receive cryotherapy would report lower pain scores as a primary outcome measure. This would result in less narcotic analgesia usage, and shorter hospital stays as secondary outcome measures.

DETAILED DESCRIPTION:
Objectives:

This study will attempt to assess the impact of cryotherapy on post-surgical inflammation and narcotic use. End-points for the study will be patient use of narcotics and pain level, regularly measured by nursing staff.

Patient Selection:

This study will accept all consecutive consenting patients who visit the Grady Hospital and Emory University urology clinics who require abdominal surgery.The study will require 55 patients, based on prior power calculations.

Registration/Randomization:

Because this study will enroll all consenting patients, no registration is required. Patients will be enrolled by their urologist during a standard visit. With consent, the urologist will direct the patient to the researcher. Patients will be randomized to either cryotherapy or no adjunctive therapy following abdominal surgery.

Therapy:

Patients in the cryotherapy study group will have ice packs placed on their abdominal wound for 24 hours following surgery.After 24 hours, patients had the option of using ice packs for as long as they wished.

Patient Assessment:

Patients will be assessed by the nursing staff as they would otherwise be assessed postsurgically.

Data Collection:

During recovery time in the hospital, nurses will monitor both groups of patients as they do all patients. As with all patients, nurses will ask about pain levels and check the amount of narcotics you require for pain control. This study will not require any additional effort on patients' part. Once they are discharged, patient participation in the study will be complete.

ELIGIBILITY:
Inclusion Criteria:

* Any open transperitoneal abdominal surgery with a midline incision

Exclusion Criteria:

* Additional surgeries required

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2008-05; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
Change in postoperative pain score | Participants will be followed for the duration of hospital stay, an average of 7 days
  Throughout the hospital stay nurses will assess patients pain levels. Patients will complete a visual analog score one hour postoperatively and then at 8am and 4 pm each day.

SECONDARY OUTCOMES:
Narcotic use | Participants will be followed for the duration of hospital stay, an average of 7 days
  Throughout the hospital stay nurses will check the amount of narcotics patients require for pain control. All narcotic use will be documented and converted to morphine equivalents using an equianalgesic table provided by the Emory University Department of Palliative Care.

OTHER OUTCOMES:
Length of hospital stay | Participants will be followed for the duration of hospital stay, an average of 7 days
  Length of hospital stay will be recorded in patient records.

CONTACTS AND LOCATIONS:
Overall Officials: Viraj Master, MD, PhD, Principal Investigator — Emory University
Locations (2):
- United States (2):
  - Grady Hospital, Atlanta, Georgia
  - Emory University, Urology Department, Atlanta, Georgia